

# Consent of an Adult to Be in a Research Study

In this form "you" means a person 18 years of age or older who is being asked to volunteer to participate in this study.

| Medical Record # |
|------------------|

| Principal Investigator: | Bhiken Naik, M.D. |
|-------------------------|---------------------------------------|
| | University of Virginia Health System. |
| | P.O. Box 800710 |
| | Charlottesville, VA 22908 |
| | Phone: 434-924-2283 |
| Financial Support: | Merck & Co. |

# What is the purpose of this form?

This form will provide you with information about this research study. You do not have to be in the study if you do not want to. You should have all your questions answered before you agree to be in this study.

Please read this form carefully. If you want to be in the study, you will need to sign this form. You will be given a signed copy of this form.

# Who is funding this study?

This study is being funded by Merck. Merck is supplying free study drug.

# Why is this research being done?

Pain control following major spine surgery is difficult to achieve. Opiates are often necessary in high doses, and may be associated with significant side effects including constipation. Alvimopan is a drug approved by the Food and Drug Administration (FDA) and is used to help the bowel recover more quickly in patients who are having bowel surgery, so that they can eat solid foods and have regular bowel movements. Alvimopan is in a class of medications called peripherally acting mu-opioid receptor antagonists. It works by protecting the bowel from the constipation effects of opioid (narcotic) medications that are used to treat pain after surgery.

The purpose of this study is to determine if the use of alvimopan in major spine surgery reduces the time to first bowel movement. By assessing the use of alvimopam in reconstructive spinal surgery patients, researchers hope to give the scientific community insight into the broader use of this drug in other surgical populations, as well as gathering information on the impact of hospital charges and overall post-operative patient satisfaction.

You are being asked to be in this study, because you are scheduled for major spine surgery and are expected to need opioid pain medication after surgery.




Up to 60 people will be in this study at UVA.

### How long will this study take?

Your participation in this study will end when you return for your 6 week surgical follow-up. Each study visit will last about **10 minutes** 

# What will happen if you are in the study?

#### SCREENING (will take about 10 minutes to complete):

Visit 1 (Day 1):

Day of Surgery:

If you agree to participate, you will sign this consent form before any study related procedures take place. Before you can start in the study, there will be a screening period. You will have tests and procedures during this time to make sure you are eligible and it is safe for you to participate. These include the following:

- Review of your medical history
- Physical exam and vital signs ( blood pressure, heart rate)
- If you are a woman of child bearing potential, you will have a urine test to determine if you are pregnant

If these tests show you are eligible, you will begin treatment on the day of surgery...

### **RANDOMIZATION and STUDY TREATMENT**

(each visit will last about 10 minutes):

You will be randomly assigned (like the flip of a coin) to 1 of 2 study treatment groups. You have an equal chance of being assigned to any one of the groups Neither you nor your doctor can choose which group you are assigned. Neither you nor your doctor will know which study group you will get until the study is done. But if your doctor needs to know, the people doing this study can find out.

**GROUP 1:** Alvimopan

**GROUP 2:** Placebo –contains no active study medication and should have no effect.

\*\*for the purpose of this study, we will refer to both alvimopan and placebo as the "study drug"

On the day of your surgery, you will be given the study drug in the form a capsule to be taken by mouth. You will then undergo your scheduled surgery.

Following surgery, you will take the study drug by mouth twice daily for up to seven days, or until the time of discharge, whichever occurs first, to a maximum of 15 doses.




You will be given a standardized pain medication after surgery that your physician may change as they see fit for your care.

As part of the research, a member of the study team will review your medical records and record information for research purposes. This will also include financial information regarding patient charges that accrue during the hospital stay.

Daily, while you are in the hospital, a member of the study team will ask you questions about your level of pain. You will also be asked questions about your when you were able to eat solid foods, time to first flatus (gas passed), time to first ambulation and bowel movements.

| Procedure | Screening | Before<br>Surgery | Daily up to 7 days or until discharge | Discharge |
|---|---|---|---|---|
| Informed Consent | Х | | | |
| Physical Exam | Χ | | | Х |
| Review current | х | х | X | х |
| Medications | | | | |
| Opiate use | Χ | | X | Х |
| Study drug | | X | Twice daily—<br>Up to 15 doses | |
| Review health related problems | | | х | Х |
| Financial information | | | | X |
| Quality of recovery<br>Questionairre | | | | X |
| Pain scores | | | x | |
| Time of first solid food intake | | | х | |
| Time to first ambulation | | | X | |
| Time to first flatus | | | Х | |
| Time to first bowel | | | Х | |
| movement | | | | |

### **End of Study Participation:**

After you have completed the study, you will no longer receive the study drug. You will be referred to your primary care provider or specialist so that they may decide is you need to resume taking the medication you were taking before enrollment.

# What are your responsibilities in the study?

You have certain responsibilities to help ensure your safety. These responsibilities are listed below:

- You must be completely truthful about your health history.
- Follow all instructions given.
- You should tell the study doctor or study staff about any changes in your health or the way you feel.
- Answer all of the study-related questions completely.




#### If you want to know about the results before the study is done:

During the study your study leader will let you know of any test results that may be important to your health. In addition, as the research moves forward, your study leader will keep you informed of any new findings that may be important for your health or may help you decide if you want to continue in the study. The final results of the research will not be known until all the information from everyone is combined and reviewed. At that time you can ask for more information about the study results.

## What are the risks of being in this study?

Risks and side effects related to Alvimopan include:

#### Likely

- Constipation
- Flatulence (gas)
- Dyspepsia ( upset stomach)

#### **Less Likely**

- Anemia (low blood count)
- Urinary retention
- Back pain
- Hypokalemia (low potassium)

The drug has shown an increase in heart attack when used long term, but no evidence of this has been seen with short-term use.

#### **Risks for women:**

Being in this study might hurt your unborn baby, so you will not be able to join or stay in the study if you are pregnant. You must use an effective method of birth control during the study. You should also not get pregnant for 30 days after your last dose of the study drug. If you have questions about birth control, please ask the study leader. If you are pregnant now, or get pregnant during the study, please tell us right away.

#### Other unexpected risks:

You may have side effects that we do not expect or know to watch for now. Call the study leader if you have any symptoms or problems.

# Could you be helped by being in this study?

You will not benefit from being in this study. However the information researchers get from this study may help others in the future.




### What are your other choices if you do not join this study?

You do not have to be in this study to be treated for your illness or condition. You can get the usual treatment even if you choose not to be in this study. The usual treatment would include:

- Have your surgery without participating in this study
- Your physician may prescribe medication to prevent or treat constipation that could possibly be alvimopan

If you are an employee of UVa your job will not be affected if you decide not to participate in this study. If you are a student at UVa, your grades will not be affected if you decide not to participate in this study.

# Will you be paid for being in this study?

You will not get any money for being in this study.

# Will being in this study cost you any money?

The following procedures/tests, which are being done for research purposes, will be provided at no cost to you or your health insurance: **Alvimopan / placebo and questionnaires, and pregnancy test ( if applicable).** 

You and/or your insurance company must pay for any tests or care given beyond what is required in this study. In addition, you and/or your health insurance may also have to pay for other drugs or treatments that are given to help you control any side effects. You will have to pay for any costs not covered by your health plan. You may be responsible for any co-payments or deductibles. You may wish to ask for an estimate of your financial costs. You may also wish to check with your insurance company before the study starts. Ask what they will cover and if they require you to get their permission before you decide to be in the study. You will be responsible for the cost of travel to come to any study visit and for any parking costs.

# What if you are hurt in this study?

If you are hurt as a result of being in this study, there are no plans to pay you for medical expenses, lost wages, disability, or discomfort. The charges for any medical treatment you receive will be billed to your insurance. You will be responsible for any amount your insurance does not cover. You do not give up any legal rights, such as seeking compensation for injury, by signing this form.

# What happens if you leave the study early?

You can change your mind about being in the study any time. You can agree to be in the study now and change your mind later. If you decide to stop, please tell us right away. You do not have to be in this study to get services you can normally get at the University of Virginia.

 Version: 05/10/2018



Even if you do not change your mind, the study leader or the sponsor of this study can take you out of the study. Some of the reasons for doing so may include

- a) Your study physician is concerned about your health
- b) Your condition gets worse
- c) The side effects of the treatment are too dangerous for you
- d) New information shows the treatment will not work or is not safe for you
- e) You do not follow your doctor's instructions
- f) The study sponsor closes the study for safety, administrative or other reasons

### How will your personal information be shared?

The UVa researchers are asking for your permission to gather, use and share information about you for this study. If you decide not to give your permission, you cannot be in this study, but you can continue to receive regular medical care at UVA.

### If you sign this form, we may collect any or all of the following information about you:

- o Personal information such as name, and date of birth
- Your health information if required for this study. This may include a review of your medical records and test results from before, during and after the study from any of your doctors or health care providers. This may include mental health care records, substance abuse records, and/or HIV/AIDS records, financial information related to this hospitalization.

#### 0

#### Who will see your private information?

- The researchers to make sure they can conduct the study the right way, observe the effects of the study and understand its results
- People or groups that oversee the study to make sure it is done correctly
- o The sponsor(s) of this study, and the people or groups it hires to help perform or review this research
- Insurance companies or other organizations that may need the information in order to pay your medical bills or other costs of your participation in the study
- People who evaluate study results, which can include sponsors and other companies that make the drug or device being studied, researchers at other sites conducting the same study, and government agencies that provide oversight such as the Food and Drug Administration (FDA) if the study is regulated by the FDA.

Some of the people outside of UVa who will see your information may not have to follow the same privacy laws that we follow. They may release your information to others, and it may no longer be protected by those laws.

The information collected from you might be published in a medical journal. This would be done in a way that protects your privacy. No one will be able to find out from the article that you were in the study.



A description of this clinical trial will be available on *http://www.ClinicalTrials.gov*, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### What if you sign the form but then decide you don't want your private information shared?

You can change your mind at any time. Your permission does not end unless you cancel it. To cancel it, please send a letter to the researchers listed on this form. Then you will no longer be in the study. The researchers will still use information about you that was collected before you ended your participation.

A copy of this consent form will be put in your medical record. (This is not the same as the record of this research study.) This means that everyone who is allowed to see your medical records will be able to find out that you are in this study. This is done so your regular doctors will know what you receive as part of this study. If you have other health problems during the study, they will be able to treat you properly.

#### Please contact the researchers listed below to:

- Obtain more information about the study
- Ask a question about the study procedures or treatments
- Report an illness, injury, or other problem (you may also need to tell your regular doctors)
- Leave the study before it is finished
- Express a concern about the study

#### **Principal Investigator:**

Bhiken Naik, M.D.
University of Virginia Health System.
P.O. Box 800710
Charlottesville, VA 22908 Phone: 434-924-2283

# What if you have a concern about this study?

You may also report a concern about this study or ask questions about your rights as a research subject by contacting the Institutional Review Board listed below.

University of Virginia Institutional Review Board for Health Sciences Research PO Box 800483 Charlottesville, Virginia 22908 Telephone: 434-924-9634

When you call or write about a concern, please give as much information as you can. Include the name of the study leader, the IRB-HSR Number (at the top of this form), and details about the problem. This will help officials look into your concern. When reporting a concern, you do not have to give your name.

 Version: 05/10/2018



# **Signatures**

# What does your signature mean?

Before you sign this form, please ask questions about any part of this study that is not clear to you. Your signature below means that you have received this information and all your questions have been answered. If you sign the form it means that you agree to join the study. You will receive a copy of this signed document.

| Consent From Adult | | |
|---|---|---|
| PARTICIPANT | PARTICIPANT | DATE |
| (SIGNATURE) To be completed by participant if | (PRINT) 18 years of age or older. | |
| | | study to the potential subject, allowed them have answered all their questions. |
| PERSON OBTAINING CONSENT<br>(SIGNATURE) | PERSON OBTAINING<br>CONSENT<br>(PRINT) | DATE |
| | dy doctor must be present fo | s blind or illiterate, an impartial witness not<br>r the consenting process and sign the<br>ipant Signature line above. |
| | ortunity to ask any questions | nted orally in my presence to the <b>identified</b> he/she had about the study. I also agree that participate in this trial. |
| Please indicate with check box th Subject | e identified individual(s): | |
| IMPARTIAL WITNESS<br>(SIGNATURE) | IMPARTIAL WITNESS (PRINT) | DATE |

